CLINICAL TRIAL: NCT00229710
Title: An Open-Label, Multi-Center, Long-Term Extension Study to Evaluate the Safety and Tolerability of Oral Tesaglitazar 0.5mg When Added to Insulin Therapy in Patients With Type 2 Diabetes Mellitus (GALLEX 9)
Brief Title: GALLEX 9: Safety and Tolerability of Oral Tesaglitazar When Added to Insulin Therapy in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6160C00049
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type II; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar

INTERVENTIONS:
Drug: Tesaglitazar — 0.5 in combination with insulin (with or without other oral antidiabetic drugs)
  Other Names: Galida

SUMMARY:
This is a 140-week open-label, multi-center long-term extension study from GALLANT 9 to monitor the safety and tolerability of oral tesaglitazar 0.5 mg and insulin in patients with type 2 diabetes during up to 140 weeks of treatment. The total duration, including treatment and follow-up, is 143 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >= 18 years of age
* Female patients: postmenopausal; hysterectomized; or, if of childbearing potential, using a reliable method of birth control.
* Completed the last two visits of the randomized treatment period in GALLANT 9

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, or neutropenia (low white blood cells)
* Creatinine levels of above twice the normal range
* Creatine kinase of above 3 times the upper limit of normal
* Previous enrollment in this long-term extension study
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram which, in the judgment of the investigator, would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2005-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Adverse events
Laboratory variables
Physical examination
Cardiac evaluation
Hypoglycemic events
Electrocardiogram
Vital signs (blood pressure and pulse)
Body weight

SECONDARY OUTCOMES:
Pharmacodynamic: fasting plasma glucose, glycosylated hemoglobin A1c
Lipid variables (triglyceride, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol [HDL-C], and non-HDL-C)
Responder rates and proportion of patients on tesaglitazar who reach pre-specified target levels for triglyceride, total cholesterol, low-density lipoprotein cholesterol, HDL-C and non-HDL-C
C-reactive protein (CRP)
Central obesity (waist circumference, hip circumference, waist/hip ratio)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (69):
- United States (69):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, La Jolla, California
  - Research Site, Northridge, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Spring Valley, California
  - Research Site, Walnut Creek, California
  - Research Site, West Hills, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Dunwoody, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Chicago Heights, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Cadillac, Michigan
  - Research Site, Richmond Heights, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, North Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Dover, New Hampshire
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Cheswick, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Roseland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Renton, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Madison, Wisconsin